CLINICAL TRIAL: NCT00617058
Title: Improving Metabolic Parameters of Antipsychotic Child Treatment With Ziprasidone, Aripiprazole, and Clozapine
Acronym: ZAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated in lieu of similar,competing large, multi-site study.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor of Psychiatry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-3110 GCRC-2529
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-11

CONDITIONS: Weight Gain
Keywords: antipsychotic; metformin; children; adolescents
MeSH Terms: conditions — Weight Gain | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): metformin, 250mg-2000 mg/day, in BID to TID doses for 26 weeks. Open, flexibly adjusted.
  Interventions: Drug: metformin
- 2 (Experimental): Healthy lifestyle intervention. Additional meeting at each psychiatric visit to review weight changes, level of physical activity and healthy eating behaviors
  Interventions: Behavioral: healthy lifestyle intervention
- 3 (No Intervention): Self-selected patients will be followed at major timepoints to assess weight and related measures.

INTERVENTIONS:
Drug: metformin — open dosed, randomly assigned flexible dose treatment with 250-2000mg/day divided BID or TID
  Other Names: Glucophage
  Arms: 1
Behavioral: healthy lifestyle intervention — additional component to regular psychiatric visits that includes monitoring of lifestyle and eating behaviors.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the relative risks and benefits of two approaches to the control of weight gain and other negative side effects in children and adolescents on 2nd generation antipsychotics (SGA):

* Healthy lifestyle instruction (nutritional and physical activity surveillance and advice) + continuation of current SGA;
* Add the diabetes drug, metformin + continuation of current SGA.

DETAILED DESCRIPTION:
The proposed pilot study is being conducted to obtain pilot data to support a grant application for a multi-site randomized controlled trial. The primary objective is to evaluate the relative risks and benefits of two approaches to the control of weight gain and other negative side effects in children and adolescents on 2nd generation antipsychotics (SGA). The critical question being addressed is: What can be done for the many youth who have gained substantial weight or developed high levels of lipids or glucose in their blood on an SGA; but due to their illness require continued treatment with an antipsychotic?

At least 40 youths (and no more than 60) age 10-17 that have gained substantial weight while taking a frequently used SGA: ziprasidone, aripiprazole or clozapine will be randomized to one of two treatments for 6 months:

* Healthy lifestyle instruction (nutritional and physical activity surveillance and advice) + continuation of current SGA;
* Add the diabetes drug, metformin + continuation of current SGA.
* Subjects may also elect to be in an observational arm that involves no intervention but the same major assessments.

Height, weight, body fat, and various blood tests indicative of general health will be collected during the 6 month trial to monitor the health benefits and safety of the interventions.

SGAs are associated with concerning degrees of weight gain and metabolic consequences. Children and adolescents, in whom SGAs are used increasingly for a wide variety of conditions, are particularly vulnerable to these side effects, which adversely affect health and longevity. It is imperative that researchers evaluate the efficacy and safety of interventions designed to prevent and treat the weight gain and metabolic problems caused by antipsychotic treatment of children. Lifestyle interventions and adjunctive medications all hold some promise of efficacy. However, it is essential that these strategies be rigorously evaluated as soon as possible in order to prevent the ongoing health consequences of SGA treatment in another generation of children with serious psychiatric illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10 to 17 years (inclusive).
* Receiving treatment with ziprasidone, aripiprazole or clozapine for the past 56 days or longer.
* Clinically stable on current treatment regimen (see Rationales below).
* Stable dose of current psychotropic co-medications for at least 30 days.
* BMI increase of > 7% within 3 months OR a > 0.5 BMI z-score increase within the past 24 months while taking olanzapine, quetiapine or risperidone, with maintenance of the threshold level of weight gain.
* Lifetime diagnosis of a schizophrenia spectrum disorder (schizophrenia, schizoaffective disorder, psychotic disorder NOS), a bipolar spectrum disorder (bipolar disorder, bipolar disorder NOS), certain mood disorders (mood disorder NOS, major depressive disorder with psychotic features), or certain disruptive/aggressive disorders (conduct disorder, intermittent explosive disorder, autism spectrum disorder with history of clinically significant levels of disruptive behaviors as defined below) using DSM-IV criteria determined by clinical interview and K-SADS-PL.
* Sexually active girls must agree to use an effective form of birth control or be abstinent.
* Principle caretaker is able to participate in study appointments as is clinically indicated.
* guardian and the child must agree (legally consent and assent) to participation.

Exclusion Criteria:

* Any medication that would significantly alter glucose, insulin or lipid levels. Prohibited medications will include, but are not limited to: insulin, steroids, topiramate, sibutramine, orlistat, metformin, amantadine, vitamin E (other than in standard multivitamins), antidiabetic drugs, HIV drugs.
* Major neurological disorder or medical illness that affects weight gain (e.g., unstable thyroid disease), requires a prohibited systemic medication or procedure (e.g., diabetes mellitus [insulin], chronic renal failure [steroids]) or that would prevent participation in physical activity in the healthy lifestyle program.
* Current active thyroid (TSH >18 microIU/ml), hepatic (2 LFTs >4x upper limits of normal), renal (serum Creatinine >1.4 mg/dL in females and serum Creatinine >1.5 mg/dL in males), cardiac, gastrointestinal, or adrenal disease.
* Fasting glucose > 125 mg/dL on two occasions indicating need for prompt treatment for diabetes.
* Child meets DSM-IV criteria for substance abuse or dependence disorder within the past month, not including tobacco abuse or dependence • Current treatment with more than one antipsychotic medication.
* Current treatment with more than 5 total psychotropic medications (i.e., 4 psychotropics plus SGA).
* Known hypersensitivity to metformin.
* Pregnant or breast feeding.
* Current or lifetime diagnosis of anorexia nervosa or bulimia nervosa.
* Significant risk for dangerousness to self or to others that makes participating inadvisable.
* Language issues that prevent child and/or parent from completing assessments or treatment.
* Ongoing or previously undisclosed child abuse requiring new department of social service intervention.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — University of North Carolina, Department of Psychiatry
Locations (1):
- University of North Carolina, Department of Psychiatry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects will be identified through referrals that the research program receives for other clinical trials involving the same age population with similar diagnoses. We also plan to access PHI to identify potential subjects and use MIM and the ISD helpdesk to complete hospital review of individuals ages 10-17 taking an antipsychotic.
Pre-assignment Details: Randomization will be completed using computer generated randomization schedules. In order to preserve adequate sample sizes in the cells, important variables such as pubertal status, concomitant valproic acid, concomitant stimulants, gender, race (Asian/Caucasian vs. Other), and ethnicity (Hispanic/Non-Hispanic) will be examined as covariates.
Groups:
- Co-Treatment With Metformin: metformin, 250mg-2000 mg/day, in BID to TID doses for 26 weeks. Open, flexibly adjusted.
  metformin : open dosed, randomly assigned flexible dose treatment with 250-2000mg/day divided BID or TID
- Healthy Lifestyle Instruction Group: Healthy lifestyle intervention. Additional meeting at each psychiatric visit to review weight changes, level of physical activity and healthy eating behaviors
  healthy lifestyle intervention : additional component to regular psychiatric visits that includes monitoring of lifestyle and eating behaviors.
- Elective Monitoring Control Group: For subjects who meet study criteria but are not interested in participating in a treatment study, this option for elective monitoring will be available. This group will be provided with psychiatric care, medication management, and weight monitoring and guidance for the duration of the study; however, subjects in this group will not receive any specific weight gain intervention.
Period: Overall Study
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age Categorical [Number; unit: participants]
  <=18 years | 1 |  |  | 1
  Between 18 and 65 years | 0 |  |  | 0
  >=65 years | 0 |  |  | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 17 |  |  | 17
Gender [Number; unit: participants]
  Female | 0 |  |  | 0
  Male | 1 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in BMI
Time Frame: 24 weeks
Population: This research study only enrolled a single study participant before the entire research study was terminated due to the start of a larger, multi-site trial evaluating similar outcome measures.
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | -2.65 |  |

2. Primary Outcome: Absolute Change in Weight
Time Frame: 24 weeks
Measure: Number; unit: lbs.
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
lbs. | -10.6 |  |

3. Primary Outcome: Percent Change in Fat Mass
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | 3.80 |  |

4. Secondary Outcome: Percent Change in Insulin Levels
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | -23.08 |  |

5. Secondary Outcome: Percent Change in Total Cholesterol
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | 2.84 |  |

6. Secondary Outcome: Percent Change in Triglycerides
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | 46.60 |  |

7. Secondary Outcome: Incidence of Metabolic Syndrome
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
participants | 0 |  |

8. Primary Outcome: Percent Change in Weight
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | -4.00 |  |

9. Secondary Outcome: Percent Change in Glucose Levels
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | -3.41 |  |

10. Secondary Outcome: Percent Change in HDL
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | 7.04 |  |

11. Secondary Outcome: Percent Change in LDL
Time Frame: 24 weeks
Measure: Number; unit: percent change
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Number analyzed (Participants) | 1 | 0 | 0
percent change | -5.74 |  |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the research study, which was a 6-month period.
Description: The study only enrolled one patient who was diagnosed with Major Depressive Disorder. The subject completed all 24 weeks of study treatment and was randomly assigned to the co-treatment with metformin arm. The single study participant began treatment at dose of 1500mg for 1 week, and then maintained dose of 2000mg for remainder of study.
Arm/Group | Co-Treatment With Metformin | Healthy Lifestyle Instruction Group | Elective Monitoring Control Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
In terms of study limitations, this research study was only able to enroll a single study participant before the trial was terminated prematurely due to study start-up for a larger, multisite effort examining similar outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No